CLINICAL TRIAL: NCT05681624
Title: Maternal Oxygen Supplementation for Intrauterine Resuscitation: a Multicenter Randomized Trial
Brief Title: Maternal Oxygen Supplementation for Intrauterine Resuscitation
Acronym: MOXY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Michigan (Other); University of Texas at Austin (Other); Women and Infants Hospital of Rhode Island (Other); Dell Children's Medical Center of Central Texas (Other); Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 202209042; R01HD108614 (NIH)
Record Dates: First submitted 2022-12-14; First posted 2023-01-12 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Fetal Distress; Fetal Hypoxia; Labor and Delivery Complication
MeSH Terms: conditions — Fetal Distress; Fetal Hypoxia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxygen (Other)
  Interventions: Other: Maternal oxygen supplementation
- Room air (Active Comparator)
  Interventions: Other: Room air

INTERVENTIONS:
Other: Maternal oxygen supplementation — Maternal oxygen supplementation 10 liters/minute via nonrebreather mask
  Arms: Oxygen
Other: Room air — Room air, no mask
  Arms: Room air

SUMMARY:
More than 80% of the 3 million women who labor and deliver each year in the United States undergo continuous electronic fetal monitoring (EFM) during labor in order to fetal hypoxia and prevent the transition to acidemia, expedited operative delivery, and/or neonatal morbidity. Category II EFM is the most commonly observed group of fetal heart rate features in labor. One common response to Category II EFM is maternal oxygen (O2) supplementation. The theoretic rationale for O2 administration is that it increases O2 transfer to a hypoxic fetus. There are conflicting national guidelines regarding O2 administration - the American College of Obstetricians and Gynecologists suggest O2 is ineffective, whereas the Association of Women's Health, Obstetric, and Neonatal Nurses recommend continued use given lack of definitive data on safety and efficacy. A recent national survey of nearly 600 Labor & Delivery providers in February 2022 revealed that 49% still use O2 . Thus, there remains equipoise on the topic and high-quality data on the safety of intrapartum O2 is needed. None of the trials to date have studied the effect of intrapartum O2 on important clinical measures of neonatal or maternal morbidity. This safety data is imperative because the field of obstetrics must hold supplemental O2 to the same rigorous standards applied to any drug used in pregnancy. Without data on these definitive outcomes, it will be challenging to implement evidence-based recommendations for supplemental O2 use on Labor & Delivery. The investigators will conduct a large, multicenter, randomized noninferiority trial of O2 supplementation versus room air in patients with Category II EFM in labor.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestation
* Gestational age>=37 weeks
* Spontaneous labor or induction of labor
* English or spanish speaking
* Planned continuous fetal monitoring

Exclusion Criteria:

* Preterm gestation
* Major fetal anomaly
* Multiple gestation
* Category III fetal monitoring at time of admission
* Maternal hypoxia <95%
* Planned or scheduled cesarean delivery Excluded from randomization if receiving nitrous oxide for analgesia at time of randomization.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2124 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of neonates meeting criteria for composite neonatal morbidity | Up to 28 days of life
  One of the following diagnoses: Neonatal death, acidemia, meconium aspiration with pulmonary hypertension, hypoglycemia, hypoxic ischemic encephalopathy ,hypothermia treatment, seizure, respiratory distress

SECONDARY OUTCOMES:
Perentage of patients with operative delivery (cesarean or operative vaginal delivery) | At delivery
Percentage of patients with operative delivery for the indication of nonreassuring fetal status | At delivery
Percentage of neonates with neonatal death | 28 days of life
Percentage of neonates with acidemia (pH<7.1) | At time of delivery
  On delivery cord gas
Percentage of neonates with meconium aspiration with pulmonary hypertension | Within 72 hours of delivery
Percentage of neonates with hypoglycemia | Within 24 hours of delivery
Percentage of neonates with hypoxic ischemic encephalopathy | Within 72 hours of delivery
Percentage of neonates with hypothermia treatment | Within 72 hours of delivery
Percentage of neonates with seizure | 28 days of life
Percentage of neonates with respiratory distress | Within 72 hours of delivery
umbilical artery base excess | At delivery
umbilical artery partial pressure oxygen | At delivery
umbilical artery partial pressure carbon dioxide | At delivery
Percentage of patients with composite maternal morbidity | Within 2 weeks of delivery
  any diagnosis of the following: postpartum hemorrhage [estimated blood loss >1000 mL]; severe perineal laceration, endometritis
Apgars at 5 and 10 minutes | At 5 and 10 minutes of neonatal life
Apgar<5 at 5 and 10 mins | At 5 and 10 minutes of neonatal life
Percentage of neonates with Neonatal Intensive care unit admission | Within 72 hours of delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will plan to share de-identified participant data and outcomes, study protocol, and analytic code via the NICHD Data and Specimen Hub (DASH).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Upon publication of primary analysis and planned secondary analyses.